CLINICAL TRIAL: NCT04692324
Title: Cerebrospinal Fluid Biomarkers for Brain Tumors
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Terry Burns, Principal Investigator, Mayo Clinic
Other Study IDs: 20-008832; R61NS122096 (NIH); NCI-2021-02765 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20-008832 (Other: Mayo Clinic in Rochester)
Record Dates: First submitted 2020-12-29; First posted 2020-12-31 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Central Nervous System Neoplasm
MeSH Terms: conditions — Central Nervous System Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cerebrospinal fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Basic science (biospecimen collection): Patients undergo collection of CSF samples via lumbar puncture at least 2 times. Patients may undergo additional collection of additional CSF samples if they choose.
  Interventions: Procedure: Biospecimen Collection; Other: Electronic Health Record Review; Other: Survey Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of CSF samples
  Other Names: Biological Sample Collection; Biospecimen Collected
Other: Electronic Health Record Review — Review of medical records
Other: Survey Administration — Ancillary studies

SUMMARY:
This study examines cerebrospinal biomarkers in patients with brain tumors. A biomarker is a measurable indicator of the severity or presence of your disease state. Collecting and storing samples of cerebrospinal fluid from patients with brain tumors to study in the laboratory may help doctors develop new strategies to better diagnose, monitor, and treat brain tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To collect cerebrospinal fluid (CSF) samples that can provide a resource to the research community for biomarker discovery in patients with gliomas.

SECONDARY OBJECTIVE:

I. Evaluate the feasibility of serial CSF sampling from patients with brain tumors for longitudinal evaluation of tumor biomarkers.

OUTLINE:

Patients undergo collection of CSF samples via lumbar puncture at least 2 times. Patients may undergo additional collection of additional CSF samples if they choose.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Any evidence of neoplasm involving the central nervous system (CNS) or its adjacent structures in contact with CSF. Such lesions may include but are not limited to intra-axial or extra-axial lesions, which could be benign, malignant or as yet undefined, involving the brain, spine, meninges, nerves, or vasculature or supporting structures
* Subjects must be 18 years of age or older

Exclusion Criteria:

* Patients who are under 18 years of age or are a member of a vulnerable population will be excluded from this study
* Pregnant women or women who may be pregnant are specifically excluded from study participation
* Exception will be granted for patients with diminished capacity to consent if a legally authorized representative is available
* Patients without clinical or radiographic evidence of a potentially neoplastic CNS lesion will be excluded
* Patients with an inability or unwillingness of individual or legal guardian/representative to give written informed consent will be excluded
* Any patient for whom a clinical contraindication exists to the intended route of CSF access will be excluded. For example, a patient with a large posterior fossa mass lesion at risk of herniation, or a patient with coagulopathy, or other contraindication to lumbar puncture would not be eligible to participate via use of lumbar puncture for CSF access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with known or suspected brain tumors
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-01-14 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Collection cerebrospinal fluid (CSF) samples that can provide a resource to the research community for biomarker discovery | Up to study completion

SECONDARY OUTCOMES:
Feasibility of serial cerebrospinal fluid (CSF) sampling | Up to study completion

CONTACTS AND LOCATIONS:
Overall Officials: Terence C. Burns, M.D., Ph.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials